CLINICAL TRIAL: NCT00485641
Title: Screening of Inpatient Rehabilitation Stroke Patients for Their Potential to Qualify to Use the Saeboflex Dynamic Hand Orthosis
Brief Title: Saeboflex Dynamic Hand Orthosis for Inpatient Rehabilitation Stroke Patients
Status: Completed | Type: Observational
Sponsor: Kessler Foundation (Other)
Collaborators: Saebo, Inc. (Industry)
Other Study IDs: E-516-05
Record Dates: First submitted 2007-06-11; First posted 2007-06-13 (Estimated); Last update posted 2007-06-13 (Estimated); Status verified 2007-06

CONDITIONS: Stroke
Keywords: Stroke; SaeboFlex; Hand function
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: SaeboFlex Dynamic Hand Orthosis
Procedure: Saebo F.T.M. Arm Training Program

SUMMARY:
The purpose of this study is to determine what the potential utility of the Functional Tone Management (F.T.M) Arm Training Program using the SaeboFlex in an inpatient stroke rehabiliation hospital

DETAILED DESCRIPTION:
Therapeutic interventions for the recovery of hand function after a neurological injury have historically been very limited. A significant body of research now supports the use of an upper extremity retraining approach for functional recovery after neurological injury. Few therapeutic approaches offer any intervention specifically focused on grasp and release retraining. In an effort to address this deficit, the SaeboFlex dynamic hand orthosis was developed by occupational therapists. The F.T.M. Arm Training Program has been safely used by hundreds of occupational and physical therapists on over one thousand patients in outpatient neurological rehabilitation over the last 2 years. It is currently an accepted modality of treatment for the management of hand paresis in the acquired brain injury outpatient population. Two factors, other than the severity of the initial injury, have been clinically identified as having a significant affect on the outcomes achieved in F.T.M. Arm Training treatment. They are learned non-use and soft tissue shortening of the finger flexors. All treatment delivered to the subjects that partake in this study will be clinical care and the only research component of this study will be the assessment of outcomes. The purpose of this study is to explore the potential patient population that may qualify to use the SaeboFlex Dynamic Hand Orthosis as a therapeutic option in the inpatient population.

ELIGIBILITY:
Inclusion Criterion:

* All patients admitted to the Stroke Rehabilitation Program at the Kessler Institute for Rehabilitation locations (East Orange, Saddlebrook, and Chester).
* Approval from treating physician.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2005-08; Study Completion 2007-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elie P Elovic, M.D., Principal Investigator — Kessler Medical Rehabilitation Research & Education Center
Locations (3):
- United States (3):
  - Kessler Institute for Rehabilitation, Chester, New Jersey
  - Kessler Institute for Rehabilitation, East Orange, New Jersey
  - Kessler Institute for Rehabilitation, Saddle Brook, New Jersey